CLINICAL TRIAL: NCT04581902
Title: Biomarkers of Depression and Treatment Response
Acronym: SUNSET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-28340
Record Dates: First submitted 2020-07-27; First posted 2020-10-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major
Keywords: transcranial magnetic stimulation; depression; biomarker; TMS; neuroimaging; rTMS
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This will be a parallel-groups, stratified interventional study to investigate methods of optimizing clinical care in patients diagnosed with MDD.
Who Masked: Outcomes Assessor
Masking Description: A third party assessor will conduct a biweekly MADRS clinician rating to assess depression symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Morning rTMS treatment (Experimental): Eligible participants will be assigned to the afternoon treatment group. Prior to the onset of rTMS treatment, EEG scans and magnetic resonance imaging (MRI) sessions including diffusion weighted imaging will be recorded as baseline measures. These measures will also be repeated at treatment midpoint and within one month of rTMS discontinuation in order to track structural and functional changes that occur over the course of treatment. Participants will complete an initial screening followed by 30-40 daily sessions of repetitive transcranial magnetic stimulation (rTMS) to the dorsolateral prefrontal cortex (DLPFC), completed with their TMS provider.
  Interventions: Device: rTMS therapy
- Afternoon rTMS treatment (Experimental): Eligible participants will be assigned to the afternoon treatment group. Prior to the onset of rTMS treatment, EEG scans and magnetic resonance imaging (MRI) sessions including diffusion weighted imaging will be recorded as baseline measures. These measures will also be repeated at treatment midpoint and within one month of rTMS discontinuation in order to track structural and functional changes that occur over the course of treatment. Participants will complete an initial screening followed by 30-40 daily sessions of repetitive transcranial magnetic stimulation (rTMS) to the dorsolateral prefrontal cortex (DLPFC), completed with their TMS provider.
  Interventions: Device: rTMS therapy

INTERVENTIONS:
Device: rTMS therapy — rTMS treatment parameters will be determined by TMS care providers. Typical TMS settings for MDD involve rTMS applied at 10 Hz with an intensity of 120 % of resting motor threshold. Forty trains of 4 s duration with 11s of trains is typically applied (3000 pulses per day), resulting in approximately 90,000 pulses in a given treatment course.
  Other Names: repetitive TMS; repetitive transcranial magnetic stimulation

SUMMARY:
This study is a stratified, parallel-group, single-center study utilizing multimodal imaging techniques to identify biomarkers for Major Depressive Disorder (MDD). The study goal is to identify biomarkers for MDD and treatment response that can be implemented in clinical diagnosis and care as valid and reliable measures, through monitoring neurophysiological and electrophysiological changes across the course of transcranial magnetic stimulation (TMS) treatment.

DETAILED DESCRIPTION:
First, the study will examine the replicability and prognostic utility of two previously identified potential biomarkers for MDD using resting state imaging. Second, investigators will conduct an exploratory, whole brain analysis combining EEG and imaging techniques to identify new potential biomarkers for MDD and treatment response as participants complete a course of TMS treatment. It is the hope to shed new light on the mechanisms underlying depression and relapse, which may allow for a more effective, personalized selection of treatment course.

Participants will complete initial screening and baseline evaluation, along with resting-state functional magnetic resonance imaging (fMRI), diffusion tensor imaging (DTI) and electroencephalography (EEG) scans prior to the initial TMS treatment. Participants will complete 30-36 TMS sessions and a post-treatment evaluation, along with mid- and post-treatment fMRI, DTI and EEG scans.

It is anticipated that participants with MDD have a specific set of neural features that can classify with high precision patients with MDD from those who do not, and that align with clinical diagnoses. This set of neural features will change across the course of treatment. Further, investigators expect that improvement as rated by a common MDD measure is modulated by time of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Meet Diagnostic and Statistical Manual-V (DSM-V) diagnostic criteria for Major Depressive Disorder in a current major depressive episode, without psychotic features.
* Has Montgomery-Asberg Depressive Rating Scale (MADRS) of > 19 at baseline, corresponding with moderate to severe depression.
* Demonstrate a moderate level of resistance to antidepressant treatment in the current episode, defined as a failure of 1-4 adequate medication trials.
* If participant is on a regimen of psychotropic medication, no changes in this regimen should be made during the period between the time at which pre-treatment and post-treatment scans are taken.
* Willing and able to undergo non-invasive brain stimulation
* Willing and able to attend research visits for approximately 8 weeks
* Willing and able to provide informed consent
* Ability to speak and read English

Exclusion Criteria:

* Diagnosed with acute or chronic psychotic symptoms of disorders (e.g. schizophrenia, schizophreniform, schizoaffective disorder) in the current depressive episode.
* Has neurological conditions including epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, having a history of repetitive or severe head trauma, or with primary or secondary tumors in the central nervous system.
* Presence of an implanted magnetic-sensitive medical device in or near the head, including but not limited to pacemaker, vagus nerve stimulator, or metal aneurysm clips or coils, staples, or stents.
* Generalized anxiety disorder as the primary DSM-V disorder during the current MDD episode.
* Meets criteria for alcohol or substance abuse or dependence (other than caffeine) in previous 6 months, as determined by the SCID
* History of seizures
* Implantable hardware not compatible with MRI or with the study
* Inability to comply with study daily visits
* Women who are pregnant, plan to become pregnant, or breast feeding
* Inability to speak and/or read English
* Inability to give consent
* Any active suicidal intent or plan during the current depressive episode, as determined by a score of 3 on Question #9 of Beck's Depression Inventory (scores reviewed daily by study team members versed in scoring clinical scales), or as by a subjective determination by a study clinician during any study visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS score from baseline to end of treatment | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  Effect size of active stimulation (mean difference in Montgomery Asberg Depression Rating Scale (MADRS) score) before and after morning and afternoon treatment course. Higher MADRS score indicates more severe depression; the overall score ranges from 0 to 60.
Change in resting state BOLD signal from baseline to end of treatment | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  Change in resting state functional magnetic resonance imaging BOLD signal before and after the active treatment period.
Change in resting state EEG from baseline to end of treatment | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  Change in resting state EEG (electroencephalogram) alpha band coherence before and after the active treatment period.
Change in white matter integrity from baseline to end of treatment | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  Change in white matter integrity as measured by diffusion tensor imaging (DTI) before and after the active treatment period.

SECONDARY OUTCOMES:
Change in Beck's Depression Inventory (BDI) score from baseline to end of treatment | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  The difference in Beck's Depression Inventory (BDI) score after TMS treatment course.Higher BDI score indicates more severe depression; the overall score ranges from 0 to 63.
Change in Patient Health Questionnaire (PHQ9) score from baseline to end of treatment | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  The difference in Patient Health Questionnaire (PHQ9) score after TMS treatment course. Higher PHQ9 score indicates more severe depression; the overall score ranges from 0 to 27.
Change in Generalized Anxiety Disorder (GAD-7) score from baseline to end of treatment | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  The difference in Generalized Anxiety Disorder (GAD-7) score after TMS treatment course. Higher GAD7 score indicates more severe depression; the overall score ranges from 0 to 21.
Change in Inventory of Depressive Symptomatology (IDS-30 self report) score from baseline to end of treatment. | Up to one month prior to initial TMS session (baseline) to within one month following the completion of TMS treatment (~ 8 weeks)
  The difference in Inventory of Depressive Symptomatology Self-Report (IDS-SR) score after TMS treatment course. Higher IDS score indicates more severe depression; the overall score ranges from 0 to 84.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No